CLINICAL TRIAL: NCT02301000
Title: Intestinal Microbiota Therapy Versus Metronidazole for Primary Clostridium Difficile Infection: a Randomized Controlled Trial
Brief Title: IMT for Primary Clostridium Difficile Infection
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow recruitment in pilot phase. A follow-up trial is launched (NCT03796650).
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Kjetil Garborg, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT CDI
Record Dates: First submitted 2014-11-18; First posted 2014-11-25 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; Intestinal microbiota therapy
MeSH Terms: conditions — Clostridium Infections | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intestinal microbiota therapy (Experimental): The patients allocated to this group will receive 60 ml of the anaerobically cultivated human intestinal microbiota through a rectal catheter.
  Interventions: Biological: Intestinal microbiota therapy
- Metronidazole (Active Comparator): The patients allocated to this group will receive metronidazole 400 mg t.i.d. for 10 days
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Biological: Intestinal microbiota therapy — 60 ml of ACHIM suspension will be administered through a rectal tube
  Other Names: Anaerobically cultivated human intestinal microbiota
  Arms: Intestinal microbiota therapy
Drug: Metronidazole — Peroral metronidazole 400 mg t.i.d. for ten days
  Arms: Metronidazole

SUMMARY:
This is a randomized controlled trial to compare the effect of a 10-day course of per oral metronidazole versus a one-time rectal instillation of an anaerobically cultivated human intestinal microbiota for the treatment of a first occurrence of Clostridium difficile infection (CDI). Recurrent CDI is common after standard antibiotic treatment. We hypothesize that the instillation of a healthy intestinal microbiota will be more effective in inducing a durable cure than metronidazole for primary CDI.

DETAILED DESCRIPTION:
Up to one third of patients with clostridium difficile infection treated with antibiotics experience recurrent or relapsing symptoms within a few weeks. Even with subsequent antibiotic treatment, multiple recurrences/relapses are frequent. Fecal microbiota transplantation (FMT) has been shown to be significantly more effective in curing recurrent CDI than repeated antibiotic treatment. In current guidelines, FMT is proposed as a treatment option after multiple recurrences/relapses of CDI. The rationale to reserve transplantation of donor feces for recurrent and difficult cases of CDI is a possible risk of pathogen transmittance and the cumbersome and costly process of finding a donor and screen for communicable disease. The effect of FMT for recurrent CDI, however, suggests that this therapy may be more effective than antibiotics in inducing a durable cure also for primary CDI.

We aim to use an anaerobically cultivated human intestinal microbiota (ACHIM) that has been extensively tested for pathogens, from a donor screened for communicable diseases, to avoid the need for a case-by-case donor screening. The term Intestinal Microbiota Therapy (IMT) will be used to describe the ACHIM treatment.

Patients with a first occurrence of CDI defined by diarrhea, as defined by the World Health Organization, and a positive stool test for toxigenic Clostridium difficile will be randomized 1:1 to either a 10-day course of metronidazole 400 mg t.i.d. or a rectal instillation of 60 ml ACHIM suspension.

Patients will be contacted on day 4 by an unblinded study investigator and on days 35 and 70 by a blinded study investigator to evaluate the treatment effect. In addition, the patients will register the frequency of bowel movements on days 1-4, 7, 14 and 21.

In the case of clinical deterioration, appropriate measures will be undertaken according to current guidelines.

A second instillation of ACHIM suspension will be considered on day 4 in the absence of clinical improvement.

The primary endpoint is the rate of primary cure from CDI and no sign of relapse/recurrence within 70 days, or persistent diarrhea that could be explained by other causes with three consecutive negative stool tests for toxigenic Clostridium difficile.

Treatment failure is defined as persistent diarrhea with a positive stool test for toxigenic Clostridium difficile.

Relapsing or recurrent CDI is defined as diarrhea and a positive stool test for toxigenic Clostridium difficile within 70 days of treatment initiation after an initial resolution of diarrhea.

Preliminary sample size is estimated from a hypothesis of a primary cure rate without recurrence within 70 days of 75 % with metronidazole vs. 87.5 % with IMT.

An interim analysis is planned after inclusion of the first 40 patients to guide the final sample size estimation.

Patients will be recruited at six hospitals in South-East Norway.

Before the start of the pilot phase, an independent data safety and monitoring board (DSMB) was established to monitor potential adverse events, and to advise the study team on the results of the pilot phase of the trial with regard to benefits and harms of the treatment, recruitment, and organization.

We recognized a slower than anticipated recruitment during the pilot phase of the trial. The slow recruitment was due to the current clinical practice of rapid initiation of antibiotic therapy by clinicians, before the trial team could ascertain eligible patients for enrolment.

After the inclusion of 20 eligible patients with concluded follow-up in January 2018, the DSMB met with the trial investigators on January 29 (2018), to discuss the results of the pilot phase. In light of the results, the DSMB recommended to start preparations for the main phase of the trial to validate the magnitude of the effects of FMT in primary CDI. Further, due to the nature of the results of the pilot and its potential implications on clinical practice, the DSMB recommended publication of the pilot data. This was also deemed necessary for adequate recruitment of the main trial.

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea as defined by the World Health Organization (passage of 3 or more loose or liquid stools (i.e. taking the shape of the receptacle or corresponding to Bristol stool chart types 5-7) per day, or more frequently than is normal for the individual, and
* Positive fecal test for toxigenic Clostridium difficile, and
* No evidence of CDI during the previous year.

Exclusion Criteria:

* Known presence of other stool pathogens known to cause diarrhea.
* Pregnancy and nursing.
* Patients with ongoing antibiotic treatment for other infections that cannot be stopped for at least 12 hours.
* Inflammatory bowel disease.
* Patients incapable of providing informed consent.
* Patients with <3 months life expectancy.
* Serious immunodeficiency caused by chemotherapy or other medication.
* Active immunocompromising disease.
* Patients unable to comply with protocol requirements.
* Patients in need of intensive care who are American Society of Anesthesiologists (ASA) Physical Status classification IV and V.
* Known hypersensitivity to Metronidazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02-22 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with cure without recurrence | 70 days
  Absence of diarrhea and no signs of recurrent CDI within 70 days

SECONDARY OUTCOMES:
Number of participants without diarrhea | 35 days
  Absence of diarrhea
Number of participants in which there was a need to change treatment | 4 days
  In the case of primary treatment failure, a change of treatment strategy will be considered according to current guidelines.

OTHER OUTCOMES:
Number of participants with adverse events related to CDI treatment | 1-70 days
  Patients will be contacted at 4, 35 and 70 days to identify any adverse events related to the treatment. Patients can contact a study representative at any time in case of suspected adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bretthauer, Ph.d., Study Chair — University of Oslo; Kjetil K Garborg, MD, Ph.d., Principal Investigator — Oslo University Hospital
Locations (7):
- Norway (7):
  - Vestre Viken HF, Bærum Hospital, Sandvika, Gjettum
  - Sørlandet Hospital HF, Kristiansand
  - Diakonhjemmet Hospital, Oslo
  - Lovisenberg sykehus, Oslo
  - Oslo University Hospital, Oslo
  - Telemark Hospital HF, Skien
  - Sykehuset i Vestfold, Tønsberg

REFERENCES:
- [Background] van Nood E, Dijkgraaf MG, Keller JJ. Duodenal infusion of feces for recurrent Clostridium difficile. N Engl J Med. 2013 May 30;368(22):2145. doi: 10.1056/NEJMc1303919. No abstract available. PMID 23718168
- [Background] Kassam Z, Lee CH, Yuan Y, Hunt RH. Fecal microbiota transplantation for Clostridium difficile infection: systematic review and meta-analysis. Am J Gastroenterol. 2013 Apr;108(4):500-8. doi: 10.1038/ajg.2013.59. Epub 2013 Mar 19. PMID 23511459
- [Background] Jorup-Ronstrom C, Hakanson A, Sandell S, Edvinsson O, Midtvedt T, Persson AK, Norin E. Fecal transplant against relapsing Clostridium difficile-associated diarrhea in 32 patients. Scand J Gastroenterol. 2012 May;47(5):548-52. doi: 10.3109/00365521.2012.672587. Epub 2012 Apr 2. PMID 22468996
- [Background] Lund-Tonnesen S, Berstad A, Schreiner A, Midtvedt T. [Clostridium difficile-associated diarrhea treated with homologous feces]. Tidsskr Nor Laegeforen. 1998 Mar 10;118(7):1027-30. Norwegian. PMID 9531822
- [Background] Garborg K, Waagsbo B, Stallemo A, Matre J, Sundoy A. Results of faecal donor instillation therapy for recurrent Clostridium difficile-associated diarrhoea. Scand J Infect Dis. 2010 Dec;42(11-12):857-61. doi: 10.3109/00365548.2010.499541. Epub 2010 Jul 22. PMID 20662620
- [Background] Midtvedt T, Norin E, Benno P, Dahlgren AL. Response to Surawicz et al. Am J Gastroenterol. 2013 Dec;108(12):1931-2. doi: 10.1038/ajg.2013.280. No abstract available. PMID 24300869